CLINICAL TRIAL: NCT05942378
Title: A Phase 1 Study to Evaluate the Efficacy and Safety of HRXG-K-1939 and Adebrelimab in Patients With Advanced Solid Tumors
Brief Title: A Study of HRXG-K-1939 and Adebrelimab in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, MD, Ph.D, Fudan University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT-HRXG-K-193
Record Dates: First submitted 2023-06-21; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRXG-K-1939 Combined with Adebrelimab (Experimental): Dose Escalation:
  HRXG-K-1939 at escalated dosages with Adebrelimab Experimental: Dose Expansion HRXG-K-1939 at recommended dose with Adebrelimab
  Interventions: Drug: HRXG-K-1939; Drug: Adebrelimab

INTERVENTIONS:
Drug: HRXG-K-1939 — HRXG-K-1939
  Other Names: HRXG-K-1939 is a mRNA cancer vaccines
Drug: Adebrelimab — Adebrelimab is a programmed death-ligand 1 antibody

SUMMARY:
This is a Phase 1, open-label study evaluating the efficacy and safety of HRXG-K-1939 in combination with Adebrelimab (anti-programmed death-ligand 1 [anti-PD-L1] antibody) in patients with advanced solid tumors. HRXG-K-1939 will be administered to patients in a dose escalation regimen to determine a recommended dose for expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed the informed consent form and complied with protocols requirements;
2. Patients with advanced solid tumors that are suitable for immunotherapy;
3. ECOG Performance Status of 0 or 1;
4. Life expectancy ≥ 12 weeks;
5. At least one measurable disease per RECIST v1.1;
6. Tumor specimen availability;
7. Adequate marrow and organ function;
8. Have resolution of toxic effects from prior therapy to Grade 1 or less (except for Grade ≤2 alopecia or neuropathy) per CTCAE v5.0;
9. Patients with fertility are willing to use an adequate method of contraception.

Exclusion Criteria:

1. Previously detected positive driver genes (EGFR, ALK, ROS1, etc.);
2. Have leptomeningeal, or actively progressing CNS metastases (patients with stable brain metastases can be enrolled);
3. Uncontrolled pleural effusion, pericardial effusion, or ascites;
4. Major surgical procedure within 28 days prior to initiation of study treatment or anticipation of need for a major surgical procedure during the course of the study;
5. Prior anti-cancer therapy (e.g., chemotherapy, radiotherapy, hormonal therapy, targeted therapy, immunotherapy, any other investigational or immunomodulatory drugs) within 21 days prior to initiation of study treatment;
6. Live-attenuated vaccination within 28 days prior to initiation of study treatment through 60 days after the end of study;
7. Systemic steroid therapy or other form of immunosuppressive therapy within 14 days prior to initiation of study treatment;
8. Any history of an immune-mediated Grade 4 adverse event or Grade 3 adverse event that resulted in permanent discontinuation;
9. Active or history of autoimmune disease;
10. Active tuberculosis or infection requiring treatment;
11. History of interstitial lung disease;
12. Allergic to research drug ingredients;
13. Prior malignancy within 5 years prior to study entry;
14. Solid organ or allogeneic bone marrow transplant;
15. HIV positive, HCV positive, HBV DNA copies ≥ 10^3;
16. Significant cardiovascular disease;
17. Other situations that are not suitable for inclusion in this study judged by investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Phase:RP2D | 9 months
  Dose Escalation Phase: Recommended Phase 2 Dose (RP2D) of HRXG-K-1939
• Dose Expansion Phase: Antigen-Specific T-cell Responses in Peripheral Blood | Baseline through 12 months after last HRXG-K-1939 dose
  • Dose Expansion Phase: Antigen-Specific T-cell Responses in Peripheral Blood

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | 12 months
  The proportion of patients who have a CR or PR, as determined by the Investigator at local site per RECIST 1.1.
Disease Control Rate (DCR) | 12 months
  The proportion of patients who have a CR or PR or SD, as determined by the Investigator at local site per RECIST 1.1.
Duration of Response (DoR) | 12 months
  Time from the date of first documented response until the date of documented progression or death in the absence of disease progression.
Progression Free Survival (PFS) | 12 months
  Time to progression as assessed by the Investigator at local site per RECIST 1.1, or death due to any cause.
Overall Survival (OS) | 24 months
  Time to death due to any cause
Adverse Events(AEs) | From consent to 90 days after the final dose of study drug
  Occurrence of Adverse Events(AEs) graded according to CTCAE v5.0
Biomarker analysis | Baseline through 12 months after last HRXG-K-1939 dose
  Serum cytokines (IL-10, IL-6, IL-2, TNF- α, IFN- γ ) Changes from baseline condition

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided